CLINICAL TRIAL: NCT01980901
Title: A Post-Market Approved (PMA) Post-Approval Study to Evaluate the Long-Term Safety and Effectiveness of the Ovation™/Ovation Prime™ Abdominal Stent Graft System
Brief Title: Post-Approval Study of the Ovation™/Ovation Prime™ Abdominal Stent Graft System
Status: Completed | Type: Observational
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Other Study IDs: 771-0010
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ovation™/Ovation Prime™ Abdominal Stent Graft System: Adult male and female patients.
  Interventions: Device: Ovation™/Ovation Prime™ Abdominal Stent Graft System

INTERVENTIONS:
Device: Ovation™/Ovation Prime™ Abdominal Stent Graft System — Single occurence permanent implant of AAA device.

SUMMARY:
The Post-Approval Study (PAS) will evaluate the "real world" data on the Ovation™/Ovation Prime™ Abdominal Stent Graft System along with the long-term data collected from the IDE cohort to monitor the long-term safety and effectiveness of the device.

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate the long term safety and effectiveness of the Ovation™/Ovation Prime™ Abdominal Stent Graft System for the endovascular treatment of infrarenal abdominal aortic aneurysms in a post-approval environment.

The clinical objective of the study is to evaluate the long term safety and effectiveness of the Ovation™/Ovation Prime™ Abdominal Stent Graft System assessed at 5 years through freedom from Aneurysm-Related Mortality.

Additionally, this study will evaluate the physician training program for modifications based on IDE and post-approval experience.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years of age.
2. Patients who are male or non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study).
3. Patient has signed an Institutional Review Board (IRB) approved Informed Consent Form.
4. Patient is considered by the treating physician to be a candidate for elective open surgical repair of the AAA (i.e., category I, II, or III per American Society of Anesthesiology (ASA) classification; refer to Appendix III: ASA Classification System). ASA category IV patients may be enrolled provided their life expectancy is greater than 1 year.
5. Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following:

   * Abdominal aortic aneurysm >5.0 cm in diameter
   * Aneurysm has increased in size by 0.5 cm in last 6 months.
   * Maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment
6. Patient has patent iliac or femoral arteries that allow endovascular access with the TriVascular Ovation/Ovation Prime Abdominal Stent Graft System.
7. Patient has a suitable non-aneurysmal proximal aortic neck length of ≥ 7 mm inferior to the most distal renal artery ostium.
8. Patient has a suitable non-aneurysmal distal iliac artery length (seal zone) of ≥10 mm. The resultant repair should preserve patency in at least one hypogastric artery.
9. Patient has a suitable non-aneurysmal proximal aortic neck luminal diameter between 16 and 30 mm.
10. Patient has suitable non-aneurysmal distal iliac luminal diameters between 8 and 20 mm.
11. Patient meets the following anatomic criteria: the distance from the most distal renal artery to most superior internal iliac artery measurement is at least 13 cm.
12. Patient has juxtarenal aortic neck angulation ≤ 60º if proximal neck is ≥10 mm and ≤ 45º if proximal neck is <10 mm. Patient must be willing to comply with all required follow-up exams.
13. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

1. Patient has a dissecting aneurysm.
2. Patient has an acutely ruptured aneurysm.
3. Patient has an acute vascular injury.
4. Patient has a need for emergent surgery.
5. Patient has a known thoracic aortic aneurysm or dissection.
6. Patient has a mycotic aneurysm or has an active systemic infection.
7. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina).
8. Patient has had a myocardial infarction (MI) and/or stroke (CVA) within the past 6 months.
9. Patient has a major surgical or interventional procedure planned ≤30 days of the AAA repair.
10. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
11. Patient has history of bleeding disorders or refuses blood transfusions.
12. Patient has dialysis dependent renal failure or baseline serum creatinine level >2.0 mg/dl
13. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
14. Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE), PEG-based polymers, fluorinated ethylene propylene (FEP) or nitinol.
15. Patient has a body habitus that would inhibit X-ray visualization of the aorta
16. Patient has a limited life expectancy of less than 1 year
17. Patient is currently participating in an investigational device or drug clinical trial.
18. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 320 subjects enrolled with an estimated 192 evaluable subjects at the fifth year from the following cohorts:
  * Available data from the 161 pivotal cohort subjects
  * All Continued Access subjects;
  * All subjects from the HDE PAS (reference H100008); and
  * A minimum of 59 subjects from de novo enrollment.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Freedom From Aneurysm-Related Mortality at 5 Years | 5 Years
  The primary endpoint of the Ovation™/Ovation Prime™ Abdominal Stent Graft System study will be determined by evaluating freedom from aneurysm-related mortality at five (5) years. This will be compared to a target performance goal.

SECONDARY OUTCOMES:
Composite Safety and Performance Endpoints | 1 Month & Annually 1 to 5 Years
  Serious Adverse Events (SAEs) within 30 days of the initial procedure and through 12 months and annually thereafter to 5 years
  At 30 days and 12 months and annually thereafter to 5 years, the following rates will be reported:
  * Mortality (AAA-related and all-cause)
  * Device patency
  * Conversion to open surgical repair
  * Endoleak
  * AAA enlargement
  * Stent Graft Migration
  * Device integrity
  * Secondary endovascular procedures
  * Aneurysm rupture

CONTACTS AND LOCATIONS:
Overall Officials: Syed Hussain, MD, Principal Investigator — Christie Clinical Vein and Vascular Center
Locations (1):
- Christie Clinical Vein and Vascular Center, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided